CLINICAL TRIAL: NCT03034629
Title: Assessing the Reliability and Influence of Timing of Exercise on Transcranial Magnetic Stimulation (TMS) Neuroplasticity Measures
Brief Title: Assessing the Stability of Transcranial Magnetic Stimulation Plasticity Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joyce Rios Gomes Osman, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20161183
Record Dates: First submitted 2017-01-16; First posted 2017-01-27 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-term aerobic exercise (Experimental): One bout of moderate intensity exercise (75% of maximal predicated heart rate).
  Interventions: Behavioral: Short-term aerobic exercise

INTERVENTIONS:
Behavioral: Short-term aerobic exercise — One bout of moderate intensity exercise (75% of maximal predicated heart rate).

SUMMARY:
The overall goal of this proposed study is to assess the reliability of plasticity measured by transcranial magnetic stimulation (TMS) interleaved with intermittent theta-burst stimulation plasticity measures and to assess the influence of an acute bout of aerobic exercise on TMS plasticity measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18-70 years old.
* Primary language is English
* Exercise clearance

Exclusion Criteria:

* Presence of cognitive, neurologic or orthopedic conditions that could affect performance of the testing and training procedures
* History of migraines
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistance epilepsy
* Any current history of psychiatric illness
* Any unstable medical condition
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the Principal Investigator and a decision about inclusion will be made based on the following:
* The subject's past medical history, drug does, history of recent medication changes or duration of treatment, and combination with other central nervous system active drugs.
* The published TMS guidelines review medications to considered with TMS (Rossi, Hallet, Rossini, Pascual-Leone, & Safety of TMS Consensus Group, 2009)
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Intracranial lesion
* Substance abuse or dependence within the past six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Change in cortical synaptic plasticity | Baseline, 1 week
  As measured via Transcranial Magnetic Stimulation (TMS) in mean motor evoked potential (MEP) amplitude

SECONDARY OUTCOMES:
Assess TMS plasticity measures on healthy individuals after an acute bout of exercise | Baseline, 3 weeks
  As measured via Transcranial Magnetic Stimulation (TMS) in mean motor evoked potential (MEP) amplitude after an acute bout of aerobic exercise

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Gomes-Osman, PT, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No